CLINICAL TRIAL: NCT02593877
Title: A Multi-centre, Prospective, Randomized Controlled Study to Compare Outcomes of Viscoelastic Haemostatic Assay (VHA)-Guided Resuscitation Versus Conventional Resuscitation Support in Haemorrhaging Trauma Patients
Brief Title: Implementing Treatment Algorithms for the Correction of Trauma Induced Coagulopathy
Acronym: iTACTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Oslo University Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Klinikum der Universität Köln (Other); Rigshospitalet, Denmark (Other); Oxford University Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 010770
Record Dates: First submitted 2015-10-15; First posted 2015-11-02 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Hemorrhage; Coagulopathy; Trauma
Keywords: Trauma; Hemostasis; Resuscitation; Coagulopathy; Transfusion
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VHA algorithm (Experimental): Massive transfusion protocol resuscitation aiming at ratio 1:1:1 of blood components (RBC 1: plasma 1: platelets 1) and VHA-guiding further resuscitation with blood products and procoagulant factors
  Interventions: Device: VHA algorithm
- Control (No Intervention): Massive transfusion protocol resuscitation aiming at ratio 1:1:1 of blood components (RBC 1: plasma 1: platelets 1) and conventional coagulation tests guiding further resuscitation with blood products and procoagulant factors

INTERVENTIONS:
Device: VHA algorithm — Analysis of more than 2,200 trauma subjects has enabled the definition of clinically-relevant VHA thresholds (i.e. ROTEM® and TEG® parameters) and patterns by which it is possible to rapidly identify coagulopathic patients and anticipate the need for massive transfusion. These threshold parameters have been defined and applied to the generation of an evidence-based targeted treatment algorithm (i.e. the Intervention)
  Arms: VHA algorithm

SUMMARY:
This trial compares the haemostatic effect of viscoelastic haemostatic assay (VHA)-guided transfusion strategy versus non-VHA guided transfusion strategy in haemorrhaging trauma patients. Half of the randomised patients will receive VHA-led management of bleeding, whilst the other half will receive massive transfusion protocol resuscitation using conventional coagulation tests.

DETAILED DESCRIPTION:
Trauma is the most frequent cause of death in persons aged under 40, with half of these deaths resulting from uncontrolled bleeding. 1 in 4 of all severely injured and shocked patients develop a clotting abnormality termed Trauma Induced Coagulopathy (TIC) within minutes of injury, which causes blood to continue being lost from the body faster than it can be stemmed. Many more injured patients will go on to develop different types of coagulopathy at different times during the course of their treatment, either as a result of their body's ongoing response to trauma or as a consequence of their clinical care. Ultimately coagulopathic patients have increased blood transfusion requirements and suffer more adverse outcomes (e.g. multi organ failure).

Current management of coagulopathic, haemorrhaging trauma patients comprises the unguided transfusion of large volumes of red blood cells and clotting product supplements. Without rapidly available and validated diagnostics, products are delivered empirically to patients blind to the type and severity of TIC they may have or indeed even if they do not have TIC. This study will compare outcomes of viscoelastic haemostatic assay (VHA)-guided resuscitation versus conventional management of critically bleeding trauma patients. The hypothesis is that goal-directed haemostatic resuscitation of coagulopathic bleeding trauma patients will yield improved outcomes and reduced blood product demand, compared to empiric massive transfusion therapy.

ELIGIBILITY:
Inclusion Criteria:

Adult trauma patients (according to local definitions) will be enrolled if they:

* Present with hemorrhagic shock at any time from the time of injury until admission to the emergency department (where shock is defined by HR>100 b/min and/or systolic BP<90 mmHg) AND activate the local massive transfusion protocol
* Randomized within 3 hours of injury and 1 hour of admission to the emergency department
* Agreement is provided on behalf of incapacitated patients by Personal Consultee or Nominated Consultee (e.g.trauma team leader)

Exclusion Criteria:

* Any inclusion criteria are not met

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects alive and free of massive transfusion | 24 hours
  Proportion of subjects at 24 hours post-admission who are alive and free of massive transfusion (i.e. received 10 or more units of red blood cells within 24 hours)

SECONDARY OUTCOMES:
6hr Mortality | 6 hours
  All-cause mortality at 6-hours post admission
24hr Mortality | 24 hours
  All-cause mortality at 24-hours post admission
28d Mortality | 28-days
  All-cause mortality at 28-days post admission
90d Mortality | 90-days
  All-cause mortality at 90-days post admission
Duration of coagulopathy | 28-days post admission
  The time spent in coagulopathic state, as defined by Prothrombin Time / International Ratio (PTr) PTr >1.2) from Admission until the point of hemostasis (itself defined as having occurred at the end of the first hour free of red cell transfusions and the treating clinicians believe primary hemostasis has been achieved).
Severity of coagulopathy | 28-days post admission
  Defined by the area under the Prothrombin Time / International Ratio (PTr) curve from Admission to the point of haemostasis (where time of hemostasis is defined as having occurred at the end of the first hour free of red cell transfusions and the treating clinicians believe primary hemostasis has been achieved).
Proportion of patients with corrected coagulopathy after first 8U RBC | 28-days post admission
  Proportion of patients with corrected coagulopathy after first 8U RBC
Time to hemostasis | 28-days post admission
  Time from Admission to the point of hemostasis (where time of hemostasis is defined as having occurred at the end of the first hour free of red cell transfusions and the treating clinicians believe primary hemostasis has been achieved).
Time spent in coagulopathic condition until haemostasis | 28-days post admission
  Time of haemostasis is defined the period from Admission to the point as having occurred at the end of the first hour free of red cell transfusions and the treating clinicians believe primary hemostasis has been achieved. Coagulopathy defined as PTr >1.2.
6hr Blood products transfused | 6 hours
  Total blood products (RBC, plasma, platelets alone and in total) transfused in first 6hours after admission
24hr Blood products transfused | 24 hours
  Total blood products (RBC, plasma, platelets alone and in total) transfused in first 24hours after admission
28d Ventilator-free days | 28 days
  Calculated by the subtracting the number of days spent on mechanical ventilation from 28.
28d ICU-free days | 28 days
  Calculated by the subtracting the number of days spent on intensive care unit from 28.
Length of stay | 28 days
  Length of stay will be recorded in days, for the total number spent in ICU and in Hospital. If the patient is in the hospital at any time point during a day, this day will be considered a hospital day.
Symptomatic thromboembolic events | 28 days
  Symptomatic venous thromboembolic events shall be recorded, as confirmed by radiology. Other thromboembolic events such as myocardial infarction and/or stroke shall be identified by standard clinical diagnostic investigation(s).
Transfusion-related complications | 28-days
  Incidence, category and severity of acute transfusion reactions will be defined according to UK SHOT (United Kingdom Serious Hazards of Transfusion)
Organ dysfunction | 28-days
  Organ dysfunction shall be measured as Sequential Organ Failure Assessment (SOFA) score from admission to day 28 or discharge
28d/discharge QoL | 28 days
  Health-Related Quality of Life (HRQoL) will be measured at 28 day post admission or upon discharge if sooner
90d QoL | 90 days
  Health-Related Quality of Life (HRQoL) will be measured at 90 day post admission

CONTACTS AND LOCATIONS:
Overall Officials: Karim Brohi, FCRS FRCA, Study Director — Queen Mary University of London, Barts Health NHS Trust; Christine Gaarder, MD, Principal Investigator — Oslo University Hospital
Locations (7):
- Copenhagen University Hospital, Copenhagen, Denmark
- Kliniken der Stadt Köln gGmbH, Cologne, Germany
- Academic Medical Centre, Amsterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- United Kingdom (3):
  - The Royal London Hospital, London, Greater London
  - Queens Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baksaas-Aasen K, Gall L, Eaglestone S, Rourke C, Juffermans NP, Goslings JC, Naess PA, van Dieren S, Ostrowski SR, Stensballe J, Maegele M, Stanworth SJ, Gaarder C, Brohi K, Johansson PI. iTACTIC - implementing Treatment Algorithms for the Correction of Trauma-Induced Coagulopathy: study protocol for a multicentre, randomised controlled trial. Trials. 2017 Oct 18;18(1):486. doi: 10.1186/s13063-017-2224-9. PMID 29047413